CLINICAL TRIAL: NCT04554966
Title: A Phase 1b Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Doses of ABBV-382 in Persons Living With HIV-1 (PLWH)
Brief Title: Study to Assess Adverse Events and How Intravenous (IV) or Subcutaneous (SC) ABBV-382 Moves Through the Body of Adult Participants With Human Immuno-Deficiency Virus (HIV-1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: M19-966
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Human Immunodeficiency Virus (HIV)
Keywords: Human Immunodeficiency Virus; HIV; HIV-1; ABBV-382
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Part A: ABBV-382 Dose A (Experimental): Participants will receive intravenous (IV) ABBV-382 dose A on Day 1.
  Interventions: Drug: ABBV-382
- Part A: ABBV-382 Dose B (Experimental): Participants will receive intravenous (IV) ABBV-382 dose B on Day 1.
  Interventions: Drug: ABBV-382
- Part B: Intravenous Cohort: ABBV-382 Dose A (Experimental): Participants will receive intravenous (IV) ABBV-382 dose A on Days 1, 29 and 57.
  Interventions: Drug: ABBV-382
- Part B: Intravenous Cohort: Placebo for ABBV-382 Dose A (Placebo Comparator): Participants will receive intravenous (IV) placebo for ABBV-382 dose A on Days 1, 29 and 57.
  Interventions: Drug: Placebo for ABBV-382
- Part B: Intravenous Cohort: ABBV-382 Dose B (Experimental): Participants will receive intravenous (IV) ABBV-382 dose B on Days 1, 29 and 57.
  Interventions: Drug: ABBV-382
- Part B: Intravenous Cohort: Placebo for ABBV-382 Dose B (Placebo Comparator): Participants will receive intravenous (IV) placebo for ABBV-382 dose B on Days 1, 29 and 57.
  Interventions: Drug: Placebo for ABBV-382
- Part B: Subcutaneous Cohort: ABBV-382 (Experimental): Participants will receive subcutaneous (SC) ABBV-382 dose C on Days 1, 29 and 57.
  Interventions: Drug: ABBV-382

INTERVENTIONS:
Drug: ABBV-382 — Intravenous (IV) infusion
  Arms: Part A: ABBV-382 Dose A; Part A: ABBV-382 Dose B; Part B: Intravenous Cohort: ABBV-382 Dose A; Part B: Intravenous Cohort: ABBV-382 Dose B
Drug: ABBV-382 — Subcutaneous (SC) injection
  Arms: Part B: Subcutaneous Cohort: ABBV-382
Drug: Placebo for ABBV-382 — Intravenous (IV) infusion
  Arms: Part B: Intravenous Cohort: Placebo for ABBV-382 Dose A; Part B: Intravenous Cohort: Placebo for ABBV-382 Dose B

SUMMARY:
Human immuno-deficiency virus (HIV) is the virus that causes Acquired Immuno-Deficiency Syndrome (AIDS). HIV infection is considered to be a chronic disease requiring lifelong therapy. This study will evaluate how safe ABBV-382 is and how it is absorbed, distributed and eliminated from the body in adult participants with HIV-1 infection.

ABBV-382 is an investigational drug being developed for the treatment of HIV-1 infection. This study takes place in 2 parts. In Part A, participants with HIV-1 and no history of combination antiretroviral therapy (cART) or who are off cART for more than 3 months will be enrolled to receive ABBV-382. In Part B, participants with no virus in their blood and on maintenance cART will be enrolled into one of the intravenous (IV) or subcutaneous (SC) groups. In the IV groups, participants will receive either placebo or ABBV-382 whereas participants in the SC group will receive ABBV-382. There is 1 in 3 chance that participants will receive placebo (no drug) in Part B IV groups. The IV group in Part B is double-blinded which means neither the study doctors nor the participants will know who will be given study drug or placebo. Around 52 adult participants with HIV-1 infection will be enrolled at approximately 21 sites across the United States, including Puerto Rico.

Participants in Part A will receive an intravenous (IV) dose of ABBV-382 on Day 1. Participants in Part B will receive an IV or SC dose of ABBV-382 or placebo on Days 1, 29 and 57.

There may be a higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, and presence of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) is >= 18.0 to <= 35.0 kg/m^2 after rounding to the tenths decimal.
* Must agree to use effective barrier protection during sexual activity for protection against Human Immunodeficiency Virus (HIV)-1 transmission through the last study visit.
* Female participants of childbearing potential must give consent to abide by contraception requirements.
* CD4+ count of >= 350 cells/μL at screening and at least once during the 48 weeks prior to screening.
* Negative screen for drugs of abuse and alcohol at screening. Participants with a positive marijuana screen may be included after evaluation by the investigator that the use would not interfere with adherence to study requirements, and that usage is not on a regular or chronic basis.
* Laboratory values must meet the acceptable criteria.

Part A participants must also have:

* Positive test result for anti-HIV antibody at screening.
* Plasma HIV-1 ribose nucleic acid (RNA) between 1,000 - 200,000 copies/mL at screening.
* Must be naive to combination antiretroviral therapy (cART) or have been off of cART for > 12 weeks or 5 half-lives of the drug (whichever is longer) prior to screening with documentation of at least one plasma HIV-1 RNA measurement greater than or equal to the lower limit of quantification (LLOQ) during the off cART period.
* Willing to hold on initiation of cART throughout the screening period and until 4 weeks after dosing.

Part B participants must also have:

* Positive test result for anti-HIV antibody at screening.
* Must have plasma HIV-1 RNA below the lower limit of quantification at screening and at least 24 weeks prior to screening. A single unconfirmed "blip" is allowed if preceded and followed by values below the lower limit of quantification.
* Must be HIV-1 infected on cART for at least 48 weeks prior to screening and on current cART regimen for at least 12 weeks prior to screening.

Exclusion Criteria:

* Female participants who are pregnant, breastfeeding, or considering becoming pregnant during the study.
* History or ongoing diagnosis of acquired immune deficiency syndrome (AIDS)-defining illness.
* History of or active immunodeficiency (other than HIV).
* Active autoimmune disease or history of autoimmune disease that has required systemic treatment.
* Clinically significant medical disorders (other than HIV-1 infection) that might expose the participant to undue risk of harm, confound study outcomes, or prevent the participant from completing the study.
* Active or suspected malignancy or history of malignancy (other than basal cell skin cancer or cervical carcinoma in situ) in the past 5 years.
* History or evidence of active tuberculosis (TB) disease or untreated latent TB infection at screening.
* No history of positive TB skin test or interferon gamma release assay (IGRA) or at screening which is considered clinically significant by the investigator. Participant with a history of a positive TB skin test or IGRA or at screening must have documentation of completion of a Centers for Disease Control and Prevention (CDC) recommended treatment course for latent TB. Any participant with suspicion for or diagnosis of active TB is excluded.
* Known psychiatric or substance abuse disorders that would interfere with adherence to study requirements.
* Currently enrolled in another interventional clinical study.
* Received immunomodulatory or immunosuppressive (including intravenous [IV]/oral [PO] steroids at any dose, but excluding steroids that are inhaled or topical) therapy within 24 weeks prior to the first dose of study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Incidence of Study Drug-Related Grade 3 or Higher Adverse Events (AEs) | Up to Day 255
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug as either "Reasonable Possibility" or "No Reasonable Possibility" and will assess the severity of each adverse event from Grade 1 (mild) to Grade 4 (potentially life-threatening).
Maximum Observed Serum Concentration (Cmax) of ABBV-382 (Part A and Part B) | Up to Day 225
  Maximum observed serum concentration (Cmax) of ABBV-382.
Time to Cmax (Tmax) of ABBV-382 (Part A and Part B) | Up to Day 225
  Time to Cmax (Tmax) of ABBV-382.
Area Under the Serum Concentration-Time Curve From Time 0 to Time of Last Measurable Concentration (AUCt) of ABBV-382 (Part A) | Up to Day 112
  Area under the serum concentration-time curve (AUC) from time 0 to the time of last measurable concentration (AUCt) of ABBV-382.
Area Under the Serum Concentration-Time Curve From Time 0 to Infinite Time (AUCinf) of ABBV-382 (Part A) | Up to Day 112
  AUC from time 0 to infinite time (AUCinf) of ABBV-382.
Terminal Phase Elimination Rate Constant (β) of ABBV-382 (Part A) | Up to Day 112
  Terminal phase elimination rate constant of ABBV-382.
Terminal Phase Elimination Half-Life (t1/2) of ABBV-382 (Part A) | Up to Day 112
  Terminal phase elimination half-life of ABBV-382.
Observed Concentration at the End of the 4-Week Dosing Interval (Ctrough) of ABBV-382 (Part B) | Up to Day 225
  Observed concentration at the end of the 4-week dosing interval (Ctrough) of ABBV-382.
AUC During the 4-Week Dosing Interval (AUCtau) of ABBV-382 (Part B) | Up to Day 225
  AUC during the 4-week dosing interval (AUCtau) of ABBV-382.
Terminal Phase Elimination Half-Life (t1/2) of ABBV-382 (Part B) | Day 57 to Day 225
  Terminal phase elimination half-life (t1/2) of ABBV-382 will be estimated after the third dose only.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (21):
- United States (19):
  - Franco Felizarta, Md /Id# 223815, Bakersfield, California
  - Ruane Clinical Research Group /ID# 224125, Los Angeles, California
  - Quest Clinical Research /ID# 223347, San Francisco, California
  - George Washington University Medical Faculty Associates /ID# 223493, Washington D.C., District of Columbia
  - Midway Immunology and Research Center /ID# 223500, Ft. Pierce, Florida
  - Orlando Immunology Center /ID# 223498, Orlando, Florida
  - St. Joseph Comprehensive Research Institute /ID# 246232, Tampa, Florida
  - Triple O Research Institute /ID# 223460, West Palm Beach, Florida
  - CenExcel iResearch LLC /ID# 225526, Decatur, Georgia
  - Infinite Clinical Trials - Morrow /ID# 225455, Morrow, Georgia
  - University of Iowa Hospitals and Clinics /ID# 224267, Iowa City, Iowa
  - Be Well Medical Center /ID# 223381, Berkley, Michigan
  - North Shore University Hospital Manhasset /ID# 223343, Manhasset, New York
  - The Christ Hospital /ID# 224871, Cincinnati, Ohio
  - Central Texas Clinical Research /ID# 223378, Austin, Texas
  - Prism Health North Texas - Oak Cliff Health Center /ID# 223237, Dallas, Texas
  - North Texas Infectious Diseases Consultants, P.A /ID# 223236, Dallas, Texas
  - The Crofoot Research Center, Inc /ID# 223383, Houston, Texas
  - Peter Shalit, M.D. /ID# 224252, Seattle, Washington
- Puerto Rico (2):
  - Ponce Medical School Foundation /ID# 224231, Ponce
  - Clinical Research Puerto Rico /ID# 223923, San Juan

IPD SHARING:
Plan to Share IPD: No